CLINICAL TRIAL: NCT02234141
Title: A Phase 2, Dose-Ranging, Randomized, Double-Blind, Placebo-Controlled Study of GS-4997 in Subjects With Pulmonary Arterial Hypertension
Brief Title: Selonsertib in Adults With Pulmonary Arterial Hypertension
Acronym: ARROW
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-357-1394; 2014-002131-34 (EudraCT Number)
Record Dates: First submitted 2014-09-02; First posted 2014-09-09 (Estimated); Results first posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-03

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — selonsertib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Selonsertib 2 mg (Experimental): Participants will receive selonsertib 2 milligrams (mg) for 24 weeks and may continue on this dose during the long-term treatment phase.
  Interventions: Drug: Selonsertib
- Selonsertib 6 mg (Experimental): Participants will receive selonsertib 6 mg for 24 weeks and may continue on this dose during the long-term treatment phase.
  Interventions: Drug: Selonsertib
- Selonsertib 18 mg (Experimental): Participants will receive selonsertib 18 mg for 24 weeks and may continue on this dose during the long-term treatment phase.
  Interventions: Drug: Selonsertib
- Placebo (Experimental): Participants will receive selonsertib placebo for 24 weeks, and may then be rerandomized 1:1:1 to selonsertib 2, 6, or 18 mg during the long-term treatment phase.
  Interventions: Drug: Placebo; Drug: Selonsertib

INTERVENTIONS:
Drug: Placebo — Tablet administered orally once daily
  Other Names: GS-4997
  Arms: Placebo
Drug: Selonsertib — Tablets administered orally once daily
  Other Names: GS-4997

SUMMARY:
The primary objective of this study is to evaluate the effect of selonsertib (GS-4997) on pulmonary vascular resistance (PVR), as measured by right heart catheterization (RHC) in adults with pulmonary arterial hypertension (PAH). The study will consist of a 24-week placebo-controlled treatment period and a long-term selonsertib treatment period. Participants completing the 24-week placebo-controlled period will be eligible to receive active treatment with selonsertib in the long-term treatment period.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of idiopathic pulmonary arterial hypertension (IPAH), heritable pulmonary arterial hypertension (HPAH), drug- and toxin-induced PAH, or PAH associated with connective tissue disease, human immunodeficiency virus (HIV) infection, or congenital heart defects (repaired greater than 1 year prior to Screening)
* Meet all of the following hemodynamic criteria by means of a screening right heart catheterization (RHC) completed prior to randomization:

  * Mean pulmonary artery pressure (mPAP) of greater than or equal to (≥) 25 millimeters of mercury (mm Hg)
  * Pulmonary vascular resistance (PVR) ≥ 400 dyne* second/centimeter^5 (dynes*sec/cm^5)
  * Pulmonary capillary wedge pressure (PCWP) or left ventricular end diastolic pressure (LVEDP) of less than or equal to (≤) 12 mm Hg if PVR ≥ 400 and less than (<) 500 dynes*sec/cm^5, or PCWP/LVEDP ≤ 15 mm Hg if PVR ≥ 500 dynes•sec/cm^5
* Be able to walk a distance of at least 100 meters
* Have World Health Organization (WHO) Functional Class II or III symptoms
* Meet the following criteria determined by pulmonary function tests completed no more than 24 weeks prior to screening, performed with or without bronchodilation:

  * Forced expiratory volume in one second (FEV1) ≥ 55 percent (%) of predicted normal
  * FEV1: forced vital capacity (FVC) ratio ≥ 0.60
* Receiving treatment with one or more drugs approved for PAH for ≥ 12 consecutive weeks and at stable dose for ≥ 8 consecutive weeks

Key Exclusion Criteria:

* Diagnosis of PAH associated with significant venous or capillary involvement (PCWP greater than [>] 15 mm Hg), pulmonary capillary hemangiomatosis, portal hypertension, or unrepaired congenital heart defects
* Pulmonary hypertension (PH) belonging to groups 2 to 5 of the 2013 NICE classification
* Left ventricular ejection fraction (LVEF) ≤ 40% or clinically significant ischemic, valvular or constrictive heart disease
* Uncontrolled hypertension (≥ 180/110 mm Hg) at Screening
* End stage renal disease (receiving peritoneal dialysis, hemodialysis, or status after renal transplantation)
* Severe liver disease (Child-Pugh Class C, with or without cirrhosis)

Individuals may be rescreened one additional time with prior notification to and approval by the sponsor.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2014-11; Primary Completion 2016-04 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (46):
- United States (24):
  - University of South Alabama Medical Center, Mobile, Alabama
  - Advanced Lung Disease Institute, Phoenix, Arizona
  - Arizona Pulmonary Specialist, Ltd, Phoenix, Arizona
  - University of Arizona Clinical and Translational Science (CATS) Research Center, Tucson, Arizona
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - LA Biomedical Research Institute Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado Cardiac and Vascular Center, Anschutz Inpatient Pavillion, Aurora, Colorado
  - The Emory Clinic, Atlanta, Georgia
  - University of Chicago Medicine, Chicago, Illinois
  - Boston University Medical Center, Boston, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Mary M. Parkes Center // University of Rochester Medical Center, Rochester, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Martha Morehouse Medical Pavilion, Columbus, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Inova Fairfax Medical Campus, Falls Church, Virginia
- Canada (5):
  - Peter Lougheed Center, Calgary, Alberta
  - Vancouver General Hospital, The Lung Centre // Vancouver Coastal Health, Vancouver General Hospital, Vancouver, British Columbia
  - Victoria Hospital - London Health Sciences Centre, London, Ontario
  - University Health Network, Toronto, Ontario
  - Institut Universitaire de caridologie et de pneumologie de Quebee (IUCPQ), Sainte-Foy, Quebec
- France (3):
  - CHU de Grenoble Clinique Universitaire de Pneumologie, Grenoble
  - CHU de Bicetre, Service de Pneumologie-Reanimation Respiratoire, Le Kremlin-Bicêtre
  - Hopital Cardiologique-CHRU Lille, Service de cardiologie, Lille
- Germany (6):
  - Universitatsklinikul Giessen und Marburg GmbH, Giessen, Hesse
  - Klinik III fur Innere Medizin, Herzzentrum Uniklinik Koln, Cologne
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinikum Leipzig, Leipzig
  - Klinik und Poliklinik fur Innere Medizin II, Universitatsklinikum Regensburg, Regensburg
- Universita "Sapienza"-Azienda Policlinico Umberto 1, Rome, Italy
- VU University Medical Center, Amsterdam, Netherlands
- Spain (3):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Doce (12) de Octubre, Madrid
- United Kingdom (3):
  - Scottish Pulmonary Vascular Unit, Golden Jubilee National Hospital, Clydebank, West Dunbartonshire
  - Royal Free Hampstead NHS Trust, London
  - Clinical Research Facility, Royal Hallamshrie Hospital, Sheffield

REFERENCES:
- [Derived] Rosenkranz S, Feldman J, McLaughlin VV, Rischard F, Lange TJ, White RJ, Peacock AJ, Gerhardt F, Ebrahimi R, Brooks G, Satler C, Frantz RP; ARROW Study Group. Selonsertib in adults with pulmonary arterial hypertension (ARROW): a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Respir Med. 2022 Jan;10(1):35-46. doi: 10.1016/S2213-2600(21)00032-1. Epub 2021 Aug 20. PMID 34425071

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America and Europe. The first participant was screened on 12 November 2014. The last study visit occurred on 13 December 2016.
Pre-assignment Details: 185 participants were screened.
Groups:
- Selonsertib 2 mg: Participants were randomized to receive selonsertib 2 mg tablet once daily for 24 weeks during the treatment phase (Period 1) and may have continued on this dosing during the long-term treatment phase (Period 2).
- Selonsertib 6 mg: Participants were randomized to receive selonsertib 6 mg tablet once daily for 24 weeks during the treatment phase (Period 1) and may have continued on this dosing during the long-term treatment phase (Period 2).
- Selonsertib 18 mg: Participants were randomized to receive selonsertib 18 mg tablet once daily for 24 weeks during the treatment phase (Period 1) and may have continued on this dosing during the long-term treatment phase (Period 2).
- Placebo: Participants were randomized received placebo tablet once daily for 24 weeks (Period 1) and may have been rerandomized 1:1:1 to selonsertib 2, 6, or 18 mg during the long-term treatment phase (Period 2).
- Placebo to Selonsertib 2 mg: Participants received placebo in Period 1 and were rerandomized to receive selonsertib 2 mg tablet once daily during the long-term treatment phase (Period 2).
- Placebo to Selonsertib 6 mg: Participants received placebo in Period 1 and were rerandomized to receive selonsertib 6 mg tablet once daily during the long-term treatment phase (Period 2).
- Placebo to Selonsertib 18 mg: Participants received placebo in Period 1 and were rerandomized to receive selonsertib 18 mg tablet once daily during the long-term treatment phase (Period 2).
Period: Treatment Period (24 Weeks)
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo | Placebo to Selonsertib 2 mg | Placebo to Selonsertib 6 mg | Placebo to Selonsertib 18 mg
Started | 39 | 38 | 37 | 37 | 0 | 0 | 0
Completed | 35 | 32 | 35 | 32 | 0 | 0 | 0
Not Completed | 4 | 6 | 2 | 5 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Investigator's discretion | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 1 | 2 | 3 | 0 | 0 | 0
Not completed — Randomized but not treated | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Long-Term Treatment Period
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo | Placebo to Selonsertib 2 mg | Placebo to Selonsertib 6 mg | Placebo to Selonsertib 18 mg
Started | 33 (2 participants who completed Period 1 did not continue into the Long-Term Treatment Phase.) | 31 (1 participant who completed the Period 1 did not continue into the Long-Term Treatment Phase.) | 33 (2 participants who completed Period 1 did not continue into the Long-Term Treatment Phase.) | 0 (Participants were rerandomized to receive selonsertib during the Long-Term Treatment Phase.) | 10 (The Placebo group was rerandomized to receive selonsertib during the Long-Term Treatment Phase.) | 12 (The Placebo group was rerandomized to receive selonsertib during the Long-Term Treatment Phase.) | 10 (The Placebo group was rerandomized to receive selonsertib during the Long-Term Treatment Phase.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 33 | 31 | 33 | 0 | 10 | 12 | 10
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Investigator's discretion | 1 | 3 | 2 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 4 | 0 | 5 | 0 | 1 | 1 | 1
Not completed — Withdrew Consent | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Study Discontinued by Sponsor | 28 | 27 | 25 | 0 | 9 | 10 | 8

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all randomized participants who received greater than or equal to (≥) 1 dose of study drug.
Groups:
- Selonsertib 2 mg: Participants received selonsertib 2 mg tablet once daily for 24 weeks during the treatment phase (Period 1).
- Selonsertib 6 mg: Participants received selonsertib 6 mg tablet once daily for 24 weeks during the treatment phase (Period 1).
- Selonsertib 18 mg: Participants received selonsertib 18 mg tablet once daily for 24 weeks during the treatment phase (Period 1).
- Placebo: Participants received placebo tablet once daily for 24 weeks (Period 1).
- Total: Total of all reporting groups
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo | Total
Number analyzed (Participants) | 39 | 37 | 37 | 37 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (13.9) | 49 (13.7) | 48 (14.1) | 55 (15.5) | 50 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 27 | 32 | 30 | 119
  Male | 9 | 10 | 5 | 7 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 3 | 2 | 16
  Not Hispanic or Latino | 31 | 31 | 32 | 35 | 129
  Unknown or Not Reported | 2 | 1 | 2 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 0 | 3
  Asian | 0 | 3 | 0 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 35 | 33 | 36 | 35 | 139
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2
World Health Organization (WHO) Functional Class [Count of Participants; unit: Participants] — Class I: no symptoms with exercise or at rest. Class II: No symptoms at rest but uncomfortable and short of breath with normal activity such as climbing a flight of stairs, grocery shopping, or making the bed. Class III: May not have symptoms at rest but activities greatly limited by shortness of breath, fatigue, or near fainting (e.g., doing normal chores around the house, have to take breaks while doing activities of daily living). Class IV: Symptoms at rest and severe symptoms with any activity. Most participants also have edema in the feet and ankles as result of right heart failure.
  Participants
    Class II | 24 | 23 | 19 | 24 | 90
    Class III | 15 | 14 | 18 | 13 | 60
6-Minute Walk Distance (6MWD) Test [Mean (Standard Deviation); unit: meters] — The 6MWD test was conducted according to the American Thoracic Society guidelines in accordance with local standard operating procedures. It measures the distance a participant is able to walk in a period of six minutes.
  meters | 452 (111.9) | 449 (85.3) | 437 (102.7) | 412 (109.3) | 437 (103.1)
N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) [Geometric Mean (Inter-Quartile Range); unit: picograms per milliliter (pg/mL)] — NT-proBNP is used to detect, diagnose, and evaluate the severity of heart failure. In general, NT-proBNP levels are higher in participants with heart failure than those who have normal heart function.
  picograms per milliliter (pg/mL) | 385 [86 to 1177] | 431 [174 to 1134] | 352 [135 to 822] | 492 [158 to 1424] | 412 [122 to 1224]
Borg Dyspnea Index (BDI) [Mean (Standard Deviation); unit: units on a scale] — Immediately following completion of the 6-minute walk test, participants were asked to assess breathlessness using the BDI score as follows: 0 = no breathlessness, 10 = extremely strong (maximal breathlessness), Any number greater than (>) 10 = Highest possible. Therefore, the minimum for BDI score was 0 and there was no upper bound.
  units on a scale | 3.5 (2.13) | 3.7 (2.41) | 3.5 (1.53) | 3.6 (1.94) | 3.6 (2.01)
Right Ventricular Fractional Area Change (RVFAC) [Mean (Standard Deviation); unit: percentage of RV area] — RVFAC is an echocardiographic assessment of right ventricular function. Population: Participants in the Safety Analysis Set with available data were analyzed.
  percentage of RV area
    number analyzed (Participants) | 37 | 36 | 34 | 33 | 140
    (all) | 34.7 (8.00) | 33.6 (9.68) | 37.3 (8.47) | 32.3 (9.59) | 34.5 (9.04)
Tricuspid Annular Plane Systolic Excursion (TAPSE) [Mean (Standard Deviation); unit: cm] — TAPSE is an echocardiographic assessment of right ventricular function. Population: Participants in the Safety Analysis Set with available data were analyzed.
  cm
    number analyzed (Participants) | 37 | 35 | 36 | 32 | 140
    (all) | 1.5 (0.31) | 1.5 (0.37) | 1.5 (0.29) | 1.5 (0.31) | 1.5 (0.32)
Mean Right Atrial Pressure (mRAP) [Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)] — mRAP is the mean blood pressure in the right atrium of the heart.
  millimeters of mercury (mm Hg) | 8 (4.3) | 9 (4.4) | 9 (4.3) | 8 (3.5) | 8 (4.2)
Mean Pulmonary Artery Pressure (mPAP) [Mean (Standard Deviation); unit: mm Hg] — mPAP is the mean blood pressure in the pulmonary artery.
  mm Hg | 53.4 (15.28) | 56.7 (10.79) | 55.0 (12.51) | 51.3 (9.94) | 54.1 (12.38)
Pulmonary Vascular Resistance (PVR) [Mean (Standard Deviation); unit: dynes*second/centimeter^5 (dyn*sec/cm^5)] — PVR is a measure of the extent to which pulmonary circulation resists cardiac output. Population: Participants in the Safety Analysis Set with available data were analyzed.
  dynes*second/centimeter^5 (dyn*sec/cm^5)
    number analyzed (Participants) | 38 | 37 | 37 | 37 | 149
    (all) | 734 (313.4) | 806 (381.2) | 809 (366.1) | 743 (268.2) | 772 (333.5)
Cardiac Index [Mean (Standard Deviation); unit: liters/minute/square meter (L/min/m^2)] — Cardiac index is the amount of blood pumped by the heart, per minute, per meter square of body surface area.
  liters/minute/square meter (L/min/m^2) | 2.87 (0.818) | 2.86 (0.679) | 2.69 (0.649) | 2.64 (0.501) | 2.77 (0.674)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pulmonary Vascular Resistance (PVR) at Week 24, as Measured by Right Heart Catheterization (RHC)
Description: PVR is a measure of the extent to which pulmonary circulation resists cardiac output. Change from Baseline was calculated as the value at Week 24 minus the value at Baseline. The Week 24 value was defined as the last assessment at or prior to Week 24.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set (all randomized participants who received ≥ 1 dose of study drug) with available data were analyzed.
Measure: Mean (Standard Error); unit: dyne*sec/cm^5
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo
Number analyzed (Participants) | 35 | 34 | 36 | 31
dyne*sec/cm^5 | 35 (35.4) | -28 (30.2) | -21 (37.9) | 6 (28.0)
Statistical Analysis 1: Comparison: Selonsertib 2 mg vs Placebo; The protocol-specified primary analysis was to compare each selonsertib dose group with the placebo group, using Wilcoxon (van Elteren) test, with respect to change from baseline in PVR at Week 24, stratifying by randomization stratum (the underlying etiology of PAH idiopathic/heritable [yes/no] and the number of background PAH therapies they were receiving {1, 2, or greater than or equal to [≥] 3}); Test type: Other — Nonparametric pairwise comparison; p = 0.214, gvE/vE — P-value was calculated using the generalized van Elteren test/van Elteren test (gvE/vE; stratified Wilcoxon rank sum test)
Statistical Analysis 2: Comparison: Selonsertib 6 mg vs Placebo; The protocol-specified primary analysis was to compare each selonsertib dose group with the placebo group, using Wilcoxon (van Elteren) test, with respect to change from baseline in PVR at Week 24, stratifying by randomization stratum (the underlying etiology of PAH idiopathic/heritable [yes/no] and the number of background PAH therapies they were receiving [1, 2, or ≥ 3]); Test type: Other — Nonparametric pairwise comparison; p = 0.270, gvE/vE — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Selonsertib 18 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Other — Nonparametric pairwise comparison; p = 0.604, gvE/vE — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline at Week 24 in Other Cardiopulmonary Hemodynamic Measures: Cardiac Index
Description: Cardiac index is the amount of blood pumped by the heart, per minute, per meter square of body surface area. Change from Baseline was calculated as the value at Week 24 minus the value at Baseline. The Week 24 value was defined as the last assessment at or prior to Week 24.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Error); unit: L/min/m^2
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo
Number analyzed (Participants) | 35 | 34 | 36 | 31
L/min/m^2 | -0.1 (0.10) | 0.1 (0.09) | 0.0 (0.09) | 0.0 (0.09)

3. Secondary Outcome: Change From Baseline at Week 24 in Other Cardiopulmonary Hemodynamic Measures: mPAP
Description: mPAP is the mean blood pressure in the pulmonary artery. Change from Baseline was calculated as the value at Week 24 minus the value at Baseline. The Week 24 value was defined as the last assessment at or prior to Week 24.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo
Number analyzed (Participants) | 36 | 34 | 36 | 31
mm Hg | 1 (1.3) | -1 (1.1) | -3 (1.4) | 0 (1.2)

4. Secondary Outcome: Change From Baseline at Week 24 in Other Cardiopulmonary Hemodynamic Measures: mRAP
Description: mRAP is the mean blood pressure in the right atrium of the heart. Change from Baseline was calculated as the value at Week 24 minus the value at Baseline. The Week 24 value was defined as the last assessment at or prior to Week 24.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo
Number analyzed (Participants) | 36 | 34 | 36 | 31
mm Hg | 1 (0.5) | 0 (0.7) | -1 (0.5) | 1 (0.5)

5. Secondary Outcome: Change From Baseline at Week 24 in Other Cardiopulmonary Hemodynamic Measures: Mixed Venous Oxygen Saturation (SVO2) (%)
Description: SVO2 is the percentage of oxygen bound to hemoglobin in blood returning to the right side of the heart. Change from Baseline was calculated as the value at Week 24 minus the value at Baseline. The Week 24 value was defined as the last assessment at or prior to Week 24.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Error); unit: percentage of oxygen saturation
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo
Number analyzed (Participants) | 36 | 34 | 35 | 31
percentage of oxygen saturation | 0.0 (0.85) | 0.1 (2.13) | 1.1 (2.07) | -2.0 (1.00)

6. Secondary Outcome: Change From Baseline at Week 24 in Other Cardiopulmonary Hemodynamic Measures: Right Ventricular Cardiac Power (RVCP)
Description: RVCP is a cardiopulmonary hemodynamic assessment. Change from Baseline was calculated as the value at Week 24 minus the value at Baseline. The Week 24 value was defined as the last assessment at or prior to Week 24.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Error); unit: watts
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo
Number analyzed (Participants) | 35 | 34 | 36 | 31
watts | -0.01 (0.026) | 0.00 (0.024) | -0.03 (0.028) | -0.01 (0.027)

7. Secondary Outcome: Change From Baseline at Week 24 in 6MWD Test
Description: The 6MWD test was conducted according to the American Thoracic Society guidelines in accordance with local standard operating procedures. It measures the distance a participant is able to walk in a period of six minutes. Change from Baseline was calculated as the value at Week 24 minus the value at Baseline. The Week 24 value was defined as the last assessment at or prior to Week 24.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Mean (Standard Error); unit: meters
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo
Number analyzed (Participants) | 39 | 37 | 37 | 37
meters | 4.7 (6.63) | 3.5 (8.27) | -15.9 (8.01) | -15.0 (8.60)

8. Secondary Outcome: Change From Baseline at Week 24 in BDI After the 6MWD Test
Description: Immediately following completion of the 6-minute walk test, participants were asked to assess breathlessness using the BDI score as follows: 0 = no breathlessness, 10 = extremely strong (maximal breathlessness), any number > 10 = Highest possible. Therefore, the minimum for BDI score was 0 and there was no upper bound. Change from Baseline was calculated as the value at Week 24 minus the value at Baseline. The Week 24 value was defined as the last assessment at or prior to Week 24.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo
Number analyzed (Participants) | 39 | 37 | 37 | 37
units on a scale | -0.1 (0.24) | 0.1 (0.26) | 0.1 (0.23) | 0.3 (0.27)

9. Secondary Outcome: Number of Participants Experiencing Change From Baseline at Week 24 in WHO Functional Class
Description: Class I: no symptoms with exercise or at rest. Class II: No symptoms at rest but uncomfortable and short of breath with normal activity such as climbing a flight of stairs, grocery shopping, or making the bed. Class III: May not have symptoms at rest but activities greatly limited by shortness of breath, fatigue, or near fainting (e.g., doing normal chores around the house, have to take breaks while doing activities of daily living). Class IV: Symptoms at rest and severe symptoms with any activity. Most participants also have edema in the feet and ankles as result of right heart failure. The Week 24 value was defined as the last assessment at or prior to Week 24.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo
Number analyzed (Participants) | 36 | 33 | 37 | 32
Participants
  Improved | 7 | 6 | 5 | 1
  Unchanged | 27 | 24 | 28 | 29
  Worsened | 2 | 3 | 4 | 2

10. Secondary Outcome: Change From Baseline at Week 24 in NT-proBNP
Description: NT-proBNP is used to detect, diagnose, and evaluate the severity of heart failure. In general, NT-proBNP levels are higher in participants with heart failure than those who have normal heart function. Change from Baseline was calculated as the value at Week 24 minus the value at Baseline. The Week 24 value was defined as the last assessment at or prior to Week 24.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Geometric Mean (Standard Error); unit: pg/mL
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo
Number analyzed (Participants) | 39 | 37 | 37 | 37
pg/mL | 1.17 (0.093) | 1.01 (0.093) | 1.01 (0.082) | 1.25 (0.103)

11. Secondary Outcome: Change From Baseline at Week 24 in Short Form (SF-36) Physical Functioning Scale
Description: Quality of life was assessed using the SF-36 questionnaire, a self-administered multi-item survey that asks 36 questions to measure functional health and well-being from the participant's point of view and consists of eight health domains (Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health) as well as 2 summary measures (Physical Health and Mental Health). Data presented are for 1 of the domains only: Physical Functioning. Scores can range from 0 to 100, with a higher score representing a higher level of functioning. Change from Baseline was calculated as the value at Week 24 minus the value at Baseline. The Week 24 value was defined as the last assessment at or prior to Week 24.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo
Number analyzed (Participants) | 37 | 35 | 36 | 36
units on a scale | 0 (0.8) | 2 (0.9) | 0 (0.8) | 0 (0.9)

12. Secondary Outcome: Change From Baseline at Week 24 in emPHasis-10 Questionnaire Score
Description: Quality of life was assessed using the emPHasis-10 questionnaire, a disease-specific self-administered 10-question questionnaire designed for routine assessment of health-related quality of life in pulmonary hypertension. Total score can range from 0 to 50, with higher scores indicating a worse quality of life. Change from Baseline was calculated as the value at Week 24 minus the value at Baseline. The Week 24 value was defined as the last assessment at or prior to Week 24.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo
Number analyzed (Participants) | 37 | 35 | 37 | 36
units on a scale | 0 (1.1) | -1 (1.2) | 1 (1.1) | -1 (1)

13. Secondary Outcome: Change From Baseline at Week 24 in Heart Rate Recovery (HRR) After the 6MWD Test
Description: HRR was assessed after the 6MWD test. The HRR was calculated as the difference between the heart rate measured immediately after completing the 6MWD test and the second heart rate measured 1 minute after the 6MWD test. Change from Baseline was calculated as the value at Week 24 minus the value at Baseline. The Week 24 value was defined as the last assessment at or prior to Week 24.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo
Number analyzed (Participants) | 39 | 37 | 37 | 37
beats per minute (bpm) | 4.0 (2.42) | 0.1 (2.52) | -3.0 (3.07) | 2.4 (2.08)

14. Secondary Outcome: Kaplan-Meier Estimate of Time to Clinical Worsening (TTCW) Evaluated in Period 1
Description: TTCW was defined as time to the first occurrence of: death (all-cause), hospitalization for worsening pulmonary arterial hypertension (PAH) (any hospitalization for worsening PAH, lung or heart/lung transplant, atrial septostomy, or initiation of continuously infused prostanoid therapy), or disease progression (defined as both > 15% decrease from baseline in 6MWD test and WHO class III or IV symptoms at two consecutive postbaseline clinic visits separated by ≥ 14 days). TTCW was evaluated using Kaplan-Meier estimates.
Time Frame: Baseline up to Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo
Number analyzed (Participants) | 39 | 37 | 37 | 37
days | NA [NA to NA] — NA = Not reached due to insufficient number of events | NA [NA to NA] — NA = Not reached due to insufficient number of events | 225.0 [225.0 to 225.0] | 178.0 [178.0 to NA] — NA = Not reached due to insufficient number of events

15. Secondary Outcome: Change From Baseline in Echocardiographic Measures of Right Ventricular Function at Week 24: TAPSE
Description: TAPSE is an echocardiographic assessment of right ventricular function. Change from Baseline was calculated as the value at Week 24 minus the value at Baseline. The Week 24 value was defined as the last assessment at or prior to Week 24.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Error); unit: cm
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo
Number analyzed (Participants) | 37 | 35 | 35 | 32
cm | 0.0 (0.04) | -0.1 (0.06) | 0.0 (0.04) | 0.0 (0.04)

16. Secondary Outcome: Change From Baseline in Echocardiographic Measures of Right Ventricular Function at Week 24: Right Ventricular Myocardial Strain (%)
Description: Right ventricular myocardial strain is an echocardiographic assessment of right ventricular function. Change from Baseline was calculated as the value at Week 24 minus the value at Baseline. The Week 24 value was defined as the last assessment at or prior to Week 24.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Error); unit: percentage of strain
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo
Number analyzed (Participants) | 29 | 28 | 26 | 24
percentage of strain | 1 (0.7) | 2 (0.6) | -1 (0.7) | 1 (0.9)

17. Secondary Outcome: Change From Baseline in Echocardiographic Measures of Right Ventricular Function at Week 24: Tricuspid Annular Peak Sys Myocard Velocity (TAS)
Description: TAS is an echocardiographic assessment of right ventricular function. Change from Baseline was calculated as the value at Week 24 minus the value at Baseline. The Week 24 value was defined as the last assessment at or prior to Week 24.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Error); unit: centimeters per second (cm/sec)
Groups:
- Selonsertib 18 mg: Participants received selonsertib18 mg tablet once daily for 24 weeks during the treatment phase (Period 1).
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo
Number analyzed (Participants) | 37 | 37 | 35 | 32
centimeters per second (cm/sec) | 1 (0.4) | 0 (0.3) | 0 (0.2) | 0 (0.4)

18. Secondary Outcome: Change From Baseline in Echocardiographic Measures of Right Ventricular Function at Week 24: Right Ventricular Tei Index (RVTI)
Description: The Tei-index is defined as the sum of the isovolumic contraction and the isovolumic relaxation time divided by ejection time, and thus incorporates elements of both systolic and diastolic phases in the assessment of global ventricular function. An increased Tei-index results from ventricular dysfunction and provides prognostic information for a variety of myocardial conditions. The RVTI is a candidate to increase the non-invasive diagnosis of PAH because it reflects the right ventricular function, is easy to assess, and can be estimated in the same session as the echocardiographic PAP. The normal value of the RVTI is 0.28 +/- 0.04. An increased RVTI is associated with either left ventricular diastolic abnormalities or pulmonary hypertension. This score has no bounds. Change from Baseline was calculated as the value at Week 24 minus the value at Baseline. The Week 24 value was defined as the last assessment at or prior to Week 24.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo
Number analyzed (Participants) | 37 | 34 | 32 | 29
units on a scale | 0.08 (0.037) | 0.05 (0.052) | 0.01 (0.021) | -0.02 (0.038)

19. Secondary Outcome: Change From Baseline in Echocardiographic Measures of Right Ventricular Function at Week 24: Right Ventricular Fractional Area Change (RVFAC)
Description: RVFAC is an echocardiographic assessment of right ventricular function. Change from Baseline was calculated as the value at Week 24 minus the value at Baseline. The Week 24 value was defined as the last assessment at or prior to Week 24.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Error); unit: percentage of RV area
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo
Number analyzed (Participants) | 37 | 36 | 33 | 33
percentage of RV area | -0.3 (1.16) | 0.0 (1.23) | -1.1 (1.25) | -0.6 (1.12)

ADVERSE EVENTS:
Time Frame: Up to 97 weeks plus 30 days
Description: Safety Analysis Set included all randomized participants who received ≥1 dose of study drug. 10, 12, and 10 participants (from Placebo Period 1 arm who were rerandomized to receive study drug) were included in selonsertib 2 mg, selonsertib 6 mg, and selonsertib 18 mg arms, respectively, for the purpose of Adverse Event (AE) data reporting.
Groups:
- Selonsertib 2 mg: Participants received selonsertib 2 mg for 24 weeks during the treatment phase (Period 1) and during the long-term treatment phase (Period 2). AEs in this reporting group include AEs that occurred in 10 participants who were rerandomized from the Placebo Period 1 group to receive selonsertib 2 mg during the long-term treatment phase.
- Selonsertib 6 mg: Participants received selonsertib 6 mg for 24 weeks during the treatment phase (Period 1) and during the long-term treatment phase (Period 2). AEs in this reporting group include AEs that occurred in 12 participants who were rerandomized from the Placebo Period 1 group to receive selonsertib 6 mg during the long-term treatment phase.
- Selonsertib 18 mg: Participants received selonsertib 18 mg for 24 weeks during the treatment phase (Period 1) and during the long-term treatment phase (Period 2). AEs in this reporting group include AEs that occurred in 10 participants who were rerandomized from the Placebo Period 1 group to receive selonsertib 18 mg during the long-term treatment phase.
- Placebo: Participants received placebo tablet once daily for 24 weeks (Period 1). AEs reported in this group only include AEs that occurred during Period 1.
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 14/49 | 17/49 | 16/47 | 7/37
Other Adverse Events (participants affected / at risk) | 43/49 | 44/49 | 44/47 | 34/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selonsertib 2 mg (N=49) | Selonsertib 6 mg (N=49) | Selonsertib 18 mg (N=47) | Placebo (N=37)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Right ventricular failure (Cardiac disorders) | 2 | 4 | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophageal achalasia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Catheter site extravasation (General disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 2 | 0 | 0
Generalised oedema (General disorders) | 1 | 0 | 0 | 0
Infusion site inflammation (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 2 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 3 | 2 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Varicella (Infections and infestations) | 1 | 0 | 0 | 0
Transplant dysfunction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 2 | 0
Transaminases increased (Investigations) | 1 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 3 | 0 | 2 | 0
Device breakage (Product Issues) | 0 | 0 | 1 | 0
Device dislocation (Product Issues) | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Aortic arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Selonsertib 2 mg (N=49) | Selonsertib 6 mg (N=49) | Selonsertib 18 mg (N=47) | Placebo (N=37)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 4 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1 | 4 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 3 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 3 | 7 | 4 | 4
Vertigo (Ear and labyrinth disorders) | 3 | 1 | 2 | 1
Dry eye (Eye disorders) | 0 | 0 | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 5 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 3 | 3
Constipation (Gastrointestinal disorders) | 2 | 1 | 9 | 1
Diarrhoea (Gastrointestinal disorders) | 9 | 15 | 14 | 5
Nausea (Gastrointestinal disorders) | 11 | 12 | 10 | 6
Vomiting (Gastrointestinal disorders) | 3 | 6 | 4 | 3
Chest pain (General disorders) | 2 | 3 | 3 | 2
Fatigue (General disorders) | 6 | 7 | 11 | 4
Oedema peripheral (General disorders) | 1 | 8 | 5 | 2
Pyrexia (General disorders) | 3 | 2 | 0 | 2
Bronchitis (Infections and infestations) | 2 | 1 | 4 | 2
Cellulitis (Infections and infestations) | 1 | 4 | 0 | 3
Gastroenteritis (Infections and infestations) | 3 | 2 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 4 | 0 | 3 | 1
Influenza (Infections and infestations) | 4 | 1 | 0 | 2
Nasopharyngitis (Infections and infestations) | 9 | 6 | 7 | 9
Pneumonia (Infections and infestations) | 2 | 4 | 1 | 1
Respiratory tract infection (Infections and infestations) | 2 | 2 | 0 | 3
Sepsis (Infections and infestations) | 0 | 0 | 0 | 2
Sinusitis (Infections and infestations) | 3 | 2 | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 7 | 13 | 7 | 3
International normalised ratio increased (Investigations) | 5 | 2 | 1 | 1
Weight decreased (Investigations) | 3 | 1 | 3 | 1
Weight increased (Investigations) | 1 | 3 | 3 | 0
White blood cell count decreased (Investigations) | 3 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 4 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 6 | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 1 | 3 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1 | 8 | 5
Pain in jaw (Musculoskeletal and connective tissue disorders) | 4 | 3 | 5 | 0
Dizziness (Nervous system disorders) | 8 | 7 | 13 | 1
Headache (Nervous system disorders) | 8 | 15 | 20 | 8
Presyncope (Nervous system disorders) | 0 | 1 | 8 | 1
Syncope (Nervous system disorders) | 1 | 2 | 2 | 2
Abnormal dreams (Psychiatric disorders) | 2 | 2 | 5 | 1
Anxiety (Psychiatric disorders) | 0 | 3 | 1 | 1
Insomnia (Psychiatric disorders) | 3 | 3 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 14 | 8 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 12 | 7 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 3 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 4 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 5 | 6 | 2
Flushing (Vascular disorders) | 1 | 4 | 4 | 0
Hypotension (Vascular disorders) | 2 | 0 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years